CLINICAL TRIAL: NCT07390409
Title: ALIGN: A Non-randomised Study Delivering Injectable Lenacapavir for HIV Prevention Within a Pre-exposure Prophylaxis (PrEP) Choice Context in Cape Town, South Africa.
Acronym: ALIGN
Status: Not yet recruiting | Type: Observational
Sponsor: Desmond Tutu HIV Foundation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Gilead Sciences (Industry); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ALIGN; INV06512 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: Lenacapavir; Pre-exposure prophylaxis; PrEP choice; Cabotegravir
MeSH Terms: interventions — lenacapavir; cabotegravir; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and dried blood spots.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Lenacapavir Injection — Lenacapavir given every 6 months for HIV prevention.
Drug: Cabotegravir (CAB) LA — CABLA given every 2 months as HIV prevention
Drug: Tenofovi-Emtricitabine (TDF/FTC) tablet — Oral PrEP (TDF/FTC) taken daily for HIV prevention

SUMMARY:
The ALIGN study will evaluate the delivery of injectable Lenacapavir (LEN), a long-acting injectable formulation for HIV pre-exposure prophylaxis (PrEP), amongst adolescents and young people (aged 15-35 years) living within the Klipfontein-Mitchell's health sub-district of Cape Town, South Africa. LEN will be offered alongside injectable Cabotegravir long-acting (CAB LA), an injectable PrEP product already approved for use in South Africa, and oral PrEP (F/TDF) modalities (including intermittent dosing where appropriate), the current standard of care (SOC) biomedical HIV prevention in South Africa. Following counselling, participants will be able to choose which PrEP product (LEN, CAB LA, or oral PrEP) to initiate, with the option to switch at any future clinical visit, and followed for 18 months. These options will be offered from two types of delivery sites, namely public health facilities and established mobile service delivery trucks, where various forms of PrEP are currently delivered as part of outreach services and ongoing research studies (FastPrEP UCT HREC nr. 713/2021 and PrEPared to Choose 567/2023).

Lenacapavir (LEN) is a novel, first-in-class, multi-stage HIV-1 capsid inhibitor with high potency and a long half-life, allowing administration by subcutaneous injection twice yearly (1). The PURPOSE 1 study, a phase 3, double-blind, randomized, controlled trial involved adolescent girls and young women in South Africa and Uganda. Purpose 1 study found that none of the participants receiving twice-yearly LEN injection acquired HIV infection (1). Purpose 2, which was conducted amongst cisgender men who have sex with men, transgender, and non-binary populations, reported two incident infections amongst 2179 LEN users. CAB LA is an alternative long-acting injectable formulation administered by intra-muscular injection every two months. CAB LA efficacy and safety was established in the HPTN 083 and HPTN 084 studies, which indicated a 66% and 88% reduction in HIV risk compared to oral PrEP users respectively. The ongoing PrEPared to Choose study, conducted by this study team, (UCT HREC 567/2023) offers CAB LA and oral PrEP products and has demonstrated the feasibility and impact of many of the PrEP choice and delivery processes put forward in this protocol. As such, this study team has extensive experience in CAB LA and oral PrEP real-world delivery.

The ALIGN study will provide one of the first real-world (outside of the clinical trial research site) evaluations of LEN delivery with the view to evaluate firstly, what implementation strategies best support LEN initiation and persistence at the level of the PrEP provider and the PrEP user, and secondly, persistence (defined as consistent, uninterrupted use as prescribed) on LEN compared to alternative injectable products and SOC oral PrEP. The proposed study will utilise a hybrid implementation study design, with co-primary implementation and clinical aims, in the form of a non-randomised, quasi-experimental trial design. Findings from this study will be used to inform the anticipated LEN rollout into public health facilities (including ANC clinics) as well as the implementation of PrEP choice service delivery in a new era of expanded biomedical HIV prevention products. The addition of LEN will build on the experiences of implementing previous long-acting PrEP products (such as injectable long-acting Cabotegravir) and will generate practical insights to inform the scale of this innovative tool while national regulatory approvals are being sought. This will include working with communities to harness their insights and answering specific questions to support effective delivery and drive uptake and effective use of injectable PrEP (LEN and CAB LA).

Study purpose:

To evaluate the delivery strategies (public health facility and community-based) and potential impact of Lenacapavir (LEN) as PrEP, on the relative persistence of up to 3700 young people (aged 15-35 years) initiating on LEN compared to an alternative injectable product (CAB LA) and oral PrEP products (standard of care).

We hypothesize that people who select injectable PrEP will be more likely to persist on PrEP when compared with people who select oral PrEP, and further that injectable LEN will show enhanced persistence compared to injectable CAB LA.

Primary study objectives:

The primary objectives of this study are to distinguish PrEP persistence patterns across different PrEP modalities (oral PrEP vs injectable CAB vs injectable LEN as PrEP) and identify successful implementation strategies that will aid the provision of PrEP choice to adolescents and young people in South Africa from two distinct delivery platforms (public health facilities and mobile services).

DETAILED DESCRIPTION:
This proposed study will utilise a hybrid implementation design (type 2, co-primary implementation and clinical aims), in the form of a non-randomised, quasi-experimental trial design. Clinically, it aims to compare persistence among participants who self-select to use an injectable (LEN vs CAB LA) or oral PrEP modality over an 18-month period. The study will also evaluate potential implementation strategies that could be used to support PrEP adoption, initiation, and persistence at the level of the PrEP provider and PrEP user.

This research study falls within the initial implementation stage, as this will be the first post-efficacy study use of LEN amongst young people in the South African setting. This study will evaluate the delivery of LEN from both public facilities (including antenatal care services) and community settings (including mobile clinics) as well as explore methods of demand creation and choice promotion counselling within the broader PrEP offerings. Sites must be willing to administer LEN and have appropriate equipment to support administration.

This research study falls within the initial implementation stage, as this will be the first post-efficacy study use of LEN amongst young people in the South African setting. This study will evaluate the delivery of LEN from both public facilities (including antenatal care services; ANC) and community settings (including mobile clinics based in the community), as well as explore methods of demand creation and choice promotion counselling within the broader PrEP offerings.

Participants will be enrolled from a general population aged 15-35 years and will aim to include people from these groups: adolescent girls and young women (AGYW, including women who trade sex); young cis-gender men including men who have sex with men, MSM); and pregnant and lactating people.

Two mobile clinics and one public health facility will be pre-selected to host the ALIGN Project . Participants accessing sexual and reproductive health services and/or ANC services at the pre-selected public health facility, including existing PrEP users coming for product refills, will be invited to enrol on the ALIGN project. If enrolled on ALIGN, they will be able to select their preferred PrEP modalities (oral or injectable) to use for the duration of the study (18 months), with product switching allowed at any subsequent visit.

The aims of the ALIGN study are as follows:

Primary aim:

1. To determine what combination of implementation strategies best achieve PrEP initiation and persistence outcomes over the short term (6 months) and the long term (18 months). Implementation aim.
2. To explore feasibility and preference for government public health clinic (including antenatal care) vs community mobile clinic injectable PrEP delivery. Implementation aim.
3. To compare persistence between PrEP modalities (injectable Len vs vs injectable CAB vs oral PrEP) longitudinally (time to non-persistence) and segmentally (total time over which biomedical coverage of HIV risk is achieved, measured at (i) 6 months and (ii) 12 months). Clinical aim.

Secondary aims:

1. To co-design (with young people and health care providers) effective counselling and demand generation strategies that inform young people's decision to use PrEP and to choose a PrEP modality. Implementation aim
2. To compare durable persistence between PrEP modalities (injectable LEN vs injectable CAB LA vs oral PrEP), measured as the total time over which biomedical coverage of HIV risk is achieved at 18 months. Clinical aim.
3. To compare adherence (number of on-time injections or self-reported adherence for oral PrEP users) between PrEP modalities at 6 months, 12 months, and 18 months. Clinical aim.
4. To describe the acceptance, preference, safety, and tolerability of LEN, determined by self-reported adverse side effects, adverse events (including intimate partner violence), and reasons for PrEP pause, discontinuation, late injection visits or product switching. Clinical and implementation aim.
5. To explore POC rapid detection 3rd and 4th generation antibody assays vs POC qualitative Gene Xpert viral loads (NAAT) to initiate PrEP in new PrEP users. Implementation and clinical aims.
6. To describe the sexual and reproductive health package and frequency of clinic visits, testing, screening, contraception use, etc. per population group in the context of long-acting injectable PrEP methods and long-acting contraception methods (including the 3 monthly DMPA-SC).. Implementation aim

Exploratory aims:

1. To assess oral loading dose adherence and, in a limited subset explore various strategies to ensure adequate loading occurs for effective pharmacokinetics at initiation. Adherence strategies include observed dosing of first oral dose and bidirectional WhatsApp messaging before and after second oral dose. Implementation Aim
2. To describe and compare HIV incidence across the two PrEP modality arms. The sample size of the study may be insufficient to allow for a formal analysis of these outcomes. Resistance testing will be conducted for all participants that seroconvert while initiated on any PrEP product. Clinical aim

This study will offer PrEP choice amongst oral PREP (up to n=700), injectable CAB (up to n=1500), or injectable LEN as PrEP (up to n=1500). Individuals in this study will be followed for 18 months, with clinical visits timed according to product refills (oral PrEP) or administration (injectable PrEP). Missed visits will be monitored and individuals will be able to "cycle back" (i.e. return following a missed visit) at any time within the duration of the project. Participants will be allowed to switch between PrEP products according to their preference throughout the study.

Adherence is defined as on-time receipt of injections within the specific study product window (within 28 days for oral PrEP, 7 days for CAB LA, within 14 days for LEN).

Persistence is defined as continuous use of product as intended. This will be measured in two ways:

1. Longitudinal view of persistence: time to meet criteria for non-persistence from baseline.

   1. Non-persistence will be defined as >28 days gap following a scheduled CAB LA injection as per pharmacy records; and as a >14 days gap following a scheduled LEN injection (injectable PrEP).
   2. This view provides insight into how long a participant will stay persistent from initial uptake only. This view will be presented through a Kaplan-Meier analysis.
2. Segmental view of persistence: total time over the study period where biomedical coverage of HIV exposure is achieved. This view provides a more holistic assessment of the level of biomedical coverage of HIV risk that can be achieved over specific time periods (6 months, 12 months, 18 months), despite variable adherence (defined as on-time attendance at injection visits as scheduled). This view will be presented through a semi-Markov multi-state model.

Both views are necessary to assess the efficacy of real-world products in real-world settings where longitudinal persistence (time to persistence) alone fails to capture dynamic PrEP use behaviour.

Various implementation strategies to support PrEP adoption, initiation, and persistence will be implemented, monitored and reported on using a RE-AIM implementation science framework.

Primary endpoints are:

(i) Time to reach any participant sample size first (either LEN arm (n=1500), oral PrEP modalities (n=700), or CAB arm (n=1500). I.e. this endpoint will be reached once any one of the arms is fully recruited, however enrolment will continue until both the CAB LA and LEN arms have reached sample size (n=1500 respectively) (ii) Proportion of participants reached within community vs facility-based settings (iii) 12 month persistence for injectable LEN vs CAB LA vs oral PrEP. (iv) Time to missed oral or injectable PrEP pick up/visit

Secondary endpoints are:

(i) 18-month durable persistence for injectable LEN vs CAB LA vs oral PrEP (ii) Time on PrEP based on any PrEP product

ELIGIBILITY:
Inclusion Criteria:

* All participants must be HIV negative at baseline

  - 15-35 years
* All participants must have a body weight ¬> 35kg at baseline
* All participants must be currently resident in the study area
* All participants must be able to provide written, informed voluntary consent to partake in the study and willing and able to receive an injectable PrEP product
* All participants must be sexually active (has had ≥ 2 intercourse encounters within the last 3 months)

Exclusion Criteria:

* Confirmed HIV-positive test result and/or signs and symptoms of an acute HIV infection

  * Unknown or indeterminate HIV-1 status at screening or enrolment.
  * Suspected or known serious infection(s), such as active tuberculosis
  * Severe hepatic impairment or renal disease
  * Allergy or hypersensitivity to any of the PrEP agents
  * Known chronic Hepatitis B infection and currently taking oral PrEP
  * Use of contraindicated medications for LEN: ergot derivatives (ergotamine, ergonovine, dihydroergotamine, methylergonovine, ergometrine), and certain anticonvulsants.
  * Concomitant Use of known enzyme-inducing or contraindicated medications including: rifampicin, rifapentine, phenytoin, phenobarbital, carbamazepine and oxcarbazepine.
  * Do not spend a reasonable amount of time in the study area as residents, for school, or work, or are otherwise unable to participate in study visits for geographical reasons, according to the site investigator
  * Medical, social or other condition that, in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
  * Current enrolment in another interventional research study that in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (as verified by registration on the South African Medical Research Council (SAMRC) biometric co-enrolment prevention system (BCEPS)).

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: People accessing the sites (mobile clinics in Cape Town, South Africa) for general sexual and reproductive health services including PrEP will be invited to consecutively enrol on the ALIGN project. If enrolled on ALIGN, they will be able to select their preferred PrEP modalities (oral PrEP, LEN or CAB LA) to use for the duration of the study (18 months).
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To compare persistence between PrEP modalities (injectable LEN vs injectable CAB LA vs oral PrEP) longitudinally (time to non-persistence) and segmentally (total time over which biomedical coverage of HIV exposure is achieved. | Measured at 6, 12 months and 18 months
  Persistence is defined as continuous use of product as intended. This will be measured in two ways:
  1. Longitudinal view of persistence: time to meet criteria for non-persistence from baseline. This view will be presented through a Kaplan-Meier analysis.
  • Non-persistence: Defined as >28 days gap in PrEP availability for daily dosing (oral PrEP); >28 days gap in scheduled CAB LA injections as per pharmacy records; and as a ≥14 days gap following a scheduled LEN injection
  * Non-persistence may also arise if a participant discontinues PrEP but then recommences PrEP within the study timeline.
  * If a participant switches to using another PrEP product (with less than 14 day gap between products), they will be considered non-persistent on that individual PrEP product but persistent on PrEP overall.
  * If a participant defers a LEN or CAB LA injection for scheduling reasons, oral may be used as a "bridge" between injections. Participants that bridge will be defined as persistent.

CONTACTS AND LOCATIONS:
Locations (1):
- DTHF Mobile Clinics, Cape Town, WC, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected through the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol will be made available in the form of a published protocol paper. High-level, de-identified operational data on PrEP use patterns will be shared with the National Department of Health on monthly basis from first enrollment to end of study in March 2028.
Access Criteria: PI and co-Is at each site will control all rights to the data and intellectual property obtained from this project. To ensure confidentiality, data shared with project team members will be blinded (i.e. delinked from identifying participant information). All data transferred between investigators will be done securely through password-protected files. High-level, de-identified operational data on PrEP use patterns will be shared with the National Department of Health as per the national reporting stationary. All pregnancies amongst participants using LEN, CAB LA or TDF/FTC and occurring during the study, along with their outcome, will be recorded and reported to SAHPRA, UCT HREC as well as the study's collaborating partners (Gilead Sciences in the case of pregnancy while using LEN) irrespective of their association with an AE or SAE. The pregnancies will be registered on the Gilead Sciences Patient Safety Database and Viiv Healthcare/ GSK.